CLINICAL TRIAL: NCT02765204
Title: A Single-dose Cross-over Study to Assess Direct and Indirect Effects of Dapagliflozin on Pancreatic Alpha and Beta Cells in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-11421; 2015-005549-30 (EudraCT Number)
Record Dates: First submitted 2016-04-14; First posted 2016-05-06 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- DS-D-DG (Experimental): The arm label indicates the order of the given treatments in this crossover designed study (DS=Dapagliflozin and Saxagliptin, D=Dapagliflozin, DG=Dapagliflozin and Glucose).
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Glucose
- DS-DG-D (Experimental): The arm label indicates the order of the given treatments in this crossover designed study (DS=Dapagliflozin and Saxagliptin, D=Dapagliflozin, DG=Dapagliflozin and Glucose).
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Glucose
- D-DG-DS (Experimental): The arm label indicates the order of the given treatments in this crossover designed study (DS=Dapagliflozin and Saxagliptin, D=Dapagliflozin, DG=Dapagliflozin and Glucose).
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Glucose
- D-DS-DG (Experimental): The arm label indicates the order of the given treatments in this crossover designed study (DS=Dapagliflozin and Saxagliptin, D=Dapagliflozin, DG=Dapagliflozin and Glucose).
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Glucose
- DG-D-DS (Experimental): The arm label indicates the order of the given treatments in this crossover designed study (DS=Dapagliflozin and Saxagliptin, D=Dapagliflozin, DG=Dapagliflozin and Glucose).
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Glucose
- DG-DS-D (Experimental): The arm label indicates the order of the given treatments in this crossover designed study (DS=Dapagliflozin and Saxagliptin, D=Dapagliflozin, DG=Dapagliflozin and Glucose).
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Glucose

INTERVENTIONS:
Drug: Dapagliflozin
Drug: Saxagliptin
Drug: Glucose

SUMMARY:
The purpose of this study is to evaluate if Dapagliflozin has direct effect on alpha cell glucagon release.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 - 75.
2. Female subjects must meet all of the following criteria:

   1. Not breastfeeding
   2. Negative pregnancy test result (human chorionic gonadotropin, beta subunit [hCG]) at Visit 0 (screening) (not applicable to hysterectomized females).
   3. If of childbearing potential (including perimenopausal women who have had a menstrual period within 1 year), must practice and be willing to continue to practice one of the following highly effective birth control methods during the entire duration of the study:

   i. Diaphragm or partner use of condom in combination with combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
   * Oral
   * Intravaginal
   * Transdermal ii. Diaphragm or partner use of condom in combination with progestogen-only hormonal contraception associated with inhibition of ovulation:
   * Oral
   * Injectable
   * Implantable iii. Placement of an intrauterine device iv. Placement of an intrauterine hormone-releasing system v. Bilateral tubal occlusion vi. Vasectomised partner (provided that the partner is the sole sexual partner of the female subject and that the vasectomised partner has received medical assessment of the surgical success) vii. Sexual abstinence (defined as refraining from heterosexual intercourse) d) Must practice appropriate birth control as stated above for 10 weeks after the last dose of study medication
3. BMI 20 - 35.
4. Clinical T2D diagnosis at least 6 months prior to enrolment.
5. Metformin treatment, with stable dose for at least 1 month.
6. HbA1c 55 - 86 mmol/mol (7,2-10 % DCCT).

Exclusion Criteria:

1. History or sign of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Clinical diagnosis of Type 1 diabetes mellitus and/or history of diabetic ketoacidosis or positive Glutamic Acid Decarboxylase Autoantibodies test (GAD antibodies test).
3. Patients treated with antipsychotics, systemic glucocorticoids, neuropsychiatric stimulants, antidepressants with sympathetic activity, beta blockers or other pharmaceuticals rendering patient unfit for study participation as judged by the investigator.
4. Patients treated with antidiabetic medications other than Metformin.
5. Patients with any other endocrine disease except substituted hypothyroidism.
6. Significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN.
7. Patients with impaired liver or kidney function (eGFR < 60).
8. Known or suspected history of significant drug abuse.
9. History of alcohol abuse or excessive intake of alcohol as judged by investigator.
10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator.
11. Plasma donation within one month of screening or any blood donation or significant blood loss (> 400 ml) during the 3 months prior to screening.
12. Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study and /or for the patients safety.
13. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
14. Judgment by the investigator that the subject should not participate in the study if considers subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucagon levels from baseline to 0.5 hour after single-dose administration of drug. | At start and 0.5 hour after the start of each intervention
  Washout period of 2-6 weeks between the interventions
Change in plasma glucagon levels from baseline to 1 hour after single-dose administration of drug. | At start and 1 hour after the start of each intervention
Change in plasma glucagon levels from baseline to 2 hours after single-dose administration of drug. | At start and 2 hours after the start of each intervention
Change in plasma glucagon levels from baseline to 3 hours after single-dose administration of drug. | At start and 3 hours after the start of each intervention
Change in plasma glucagon levels from baseline to 5 hours after single-dose administration of drug. | At start and 5 hours after the start of each intervention
Change in plasma glucagon levels from baseline to 5.5 hours after single-dose administration of drug. | At start and 5.5 hours after the start of each intervention
Change in plasma glucagon levels from baseline to 6 hours after single-dose administration of drug. | At start and 6 hours after the start of each intervention
Change in plasma glucagon levels from baseline to 7 hours after single-dose administration of drug. | At start and 7 hours after the start of each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jan W Eriksson, MD PhD, Principal Investigator — Uppsala University
Locations (1):
- Dept of Medical Sciences Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Lundkvist P, Pereira MJ, Kamble PG, Katsogiannos P, Langkilde AM, Esterline R, Johnsson E, Eriksson JW. Glucagon Levels During Short-Term SGLT2 Inhibition Are Largely Regulated by Glucose Changes in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2019 Jan 1;104(1):193-201. doi: 10.1210/jc.2018-00969. PMID 30137410